CLINICAL TRIAL: NCT04461028
Title: The Effect of Liposomal Bupivacaine on the Quality of Recovery in Patients Undergoing Shoulder Arthroscopy
Brief Title: Liposomal Bupivacaine in Shoulder Arthroscopy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI departed from the institution and study was closed.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Nabil Elkassabany, Physician, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 832346
Record Dates: First submitted 2019-10-11; First posted 2020-07-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Randomization between Group 1 and Group 2
Who Masked: Participant, Outcomes Assessor
Masking Description: The research assistant collecting the data as well the patient will be blinded to the nature of the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GROUP 1 Liposomal Bupivacaine (Other): Will receive a 20 ml mixture of 10 ml of Liposomal Bupivacaine 1.3% and 10 ml of Bupivacaine HCl 0.5%.
  Interventions: Drug: Liposomal bupivacaine
- GROUP 2 Bupivacaine with dexamethasone (Other): Will receive 20 ml of Bupivacaine HCl 0.5% with 4 mg of preservative-free dexamethasone.
  Interventions: Drug: Bupivacaine with Dexamethasone Solution

INTERVENTIONS:
Drug: Liposomal bupivacaine — 20 ml mixture of 10 ml of Liposomal Bupivacaine 1.3% and 10 ml of Bupivacaine HCl 0.5%.
  Other Names: Exparel
  Arms: GROUP 1 Liposomal Bupivacaine
Drug: Bupivacaine with Dexamethasone Solution — 20 ml of Bupivacaine HCl 0.5% with 4 mg of preservative-free dexamethasone.
  Arms: GROUP 2 Bupivacaine with dexamethasone

SUMMARY:
Background:

The research study is being conducted to see if using the liposomal Bupivacaine for the Interscalene block will improve the patient pain control and the whole patient's experience 48 hours after surgery when compared to using the regular Marcaine (bupivacaine hydrochloride) in addition to the dexamethasone.

All preoperative, surgical, post-operative care in the recovery room, and discharge instructions will be the same as any other patient undergoing this surgery.

Study procedures:

1. After obtaining informed consent, an anesthesiologist will receive an envelope with result of randomization. Patients will receive a single injection interscalene nerve block prior to surgery
2. Patients will be randomized to one of two groups:

   * GROUP 1 liposomal Bupivacaine - will receive a 20 ml mixture of 10 ml of Liposomal Bupivacaine 1.3% and 10 ml of Bupivacaine HCl 0.5%.
   * GROUP 2 Bupivacaine with dexamethasone - will receive 20 ml of Bupivacaine HCl 0.5% with 4 mg of preservative-free dexamethasone.

4. Patients will undergo general endotracheal anesthesia with inhaled anesthetic (Sevoflurane) for a goal MAC 1.0. Other than the aforementioned interscalene nerve block, patients will not receive any other local anesthetic.

5. Patients will receive a multimodal analgesic and antiemetic regimen standardized for shoulder arthroscopies at our institution. Preoperatively, all patients will receive 300 mg of gabapentin and 1,000 mg of acetaminophen orally. Intraoperatively, patients will receive 4 mg of ondansetron and 15 mg of ketorolac intravenously. Postoperatively, patients will remain on an oral regimen of 300 mg of gabapentin three times daily for one week, and 1,000 mg of acetaminophen and 10 mg of ketorolac every 8 hours for 48 hours after surgery.

6. Additional intraoperative or postoperative opioid analgesics will be administered as needed. Patients with a history of PONV or otherwise deemed high risk for PONV by the attending anesthesiologist will receive a scopolamine patch before induction of general anesthesia.

DETAILED DESCRIPTION:
Background:

Shoulder arthroscopy is one of the most commonly performed ambulatory orthopedic procedures in the United States. However, despite advances in arthroscopic technique, significant postoperative pain remains a major challenge in the perioperative period. Regional anesthesia has played a key part in alleviating postoperative pain, particularly the use of single-shot interscalene nerve blocks. However, single-shot blocks are limited by their relatively short duration of action. The use of continuous peripheral nerve catheters is often limited by institutional resources.

As such, adjuvants can be added to the local anesthetic solution to help prolong the single-shot block. Whereas a long-acting local anesthetic such as Bupivacaine HCl can provide analgesia for 8-12 hours when deposited perineurally, the addition of adjuvants such as 4 mg preservative-free dexamethasone has been shown to prolong blocks for up to 24 hours.

Liposomal Bupivacaine (Exparel®, Pacira Pharmaceuticals, Parsippany, NJ) is a novel formulation of Bupivacaine that was approved for interscalene nerve blocks in April 2018.8 By incorporating Bupivacaine within a multivesicular liposomal suspension (DepoFoam®) that causes a slow release of the drug, it is purported to extend a nerve block's analgesic effect to at least 72 hours.9 10 ml of Liposomal Bupivacaine 1.3% (133 mg) is recommended for interscalene blocks; this solution is also often mixed with Bupivacaine HCl to complement early analgesia.

To our knowledge, no study has evaluated the effect of Liposomal Bupivacaine in the context of postoperative quality of recovery. Given the well-known postoperative pain and functional limitations of shoulder arthroscopy, the postoperative Quality of Recovery (QoR) scale is an appropriate tool to capture these outcomes. This scale assesses patient recovery in multiple domains, including physiological, nociceptive, activities of daily living, cognition and patient satisfaction. To date, the QoR scale has been used in over 100 perioperative studies and has been repeatedly validated in the postoperative setting, including ambulatory orthopedic procedures. As they have been validated over the years, the QoR has been correlated to quality of life and patient satisfaction with pain management after surgery, two key components of a successful ambulatory procedure.

Therefore, we propose a prospective randomized controlled clinical trial aiming to evaluate the effect of Liposomal Bupivacaine in this context. We hypothesize that using Liposomal Bupivacaine will improve the quality of recovery in patients undergoing shoulder arthroscopy for rotator cuff repair when compared to using Bupivicaine HCl 0.5% with preservative-free dexamethasone.

Study Objectives:

We seek to determine if Liposomal Bupivacaine 1.3% will improve the quality of recovery, as measured by QoR-15 scores, in patients undergoing shoulder arthroscopy for rotator cuff repair when compared to Bupivacaine HCl 0.5% with 4 mg of preservative-free dexamethasone as an additive.

Primary Outcome:

The primary outcome will be defined as the QoR-15 score at 48 hours after surgery.

Secondary Outcomes:

Secondary outcomes will include QoR-15 scores at 24 hours and 1 week after surgery, patient reported pain scores and opioid use at 24, 48, and 72 hours after surgery, PACU length of stay, and PACU opioids and antiemetics given.

Methods:

Study Design:

This is a prospective, randomized, controlled blinded clinical trial with a parallel design and an allocation ratio of 1:1 for the treatment groups.

Recruitment:

Patients will be identified from the surgical schedule the day before surgery and will be contacted by one of the study investigators to scan for eligibility for enrollment.

Patients will be consented the morning of their surgery by one of the study investigators or the research coordinator. Study aims and procedures will be explained to patients and all questions will be answered. There is no formal recruitment script, but the informed consent form will be carefully reviewed with the patient to ensure adequate comprehension.

Randomization:

A computer-generated randomization table will be used for patient allocation to one of the two study groups; either the Liposomal Bupivacaine group or the Bupivacaine HCl with dexamethasone group. Randomization will be done in blocks of 10 patients each.

Study procedures:

After obtaining informed consent, patients will receive a single injection interscalene nerve block prior to surgery. Patients will be randomized to one of two groups: the Liposomal Bupivacaine or Bupivacaine with dexamethasone groups. The Liposomal Bupivacaine group will receive a 20 ml mixture of 10 ml of Liposomal Bupivacaine 1.3% and 10 ml of Bupivacaine HCl 0.5%. The Bupivacaine with dexamethasone group will receive 20 ml of Bupivacaine HCl 0.2% with 4 mg of preservative-free dexamethasone. The research assistant collecting the data as well the patient will be blinded to the nature of the group assignments.

Prior to the nerve block, a block time out will be performed according to standard operating procedures with the attending anesthesiologist present. Patients will be monitored during block performance with standard ASA monitors. All patients will receive 2 L of continuous oxygen via nasal cannula. 1-2 mg midazolam will be titrated to sedative effect. All blocks will be done under ultrasound guidance using Sonosite S (Bothell, WA) machines with a high frequency linear probe (6-13 MHz). The block will be performed with strict adherence to sterile technique. After an optimal interscalene "stop-sign" view is obtained, a 21-guage needle will be inserted in-plane and the local anesthetic will be deposited with a focus on the C5 nerve root.

Patients will then undergo general endotracheal anesthesia with inhaled anesthetic (Sevoflurane) for a goal MAC 1.0. Other than the aforementioned interscalene nerve block, patients will not receive any other local anesthetic. Patients will receive a multimodal analgesic and antiemetic regimen standardized for these surgeries at this institution.

Preoperatively, all patients will receive 300 mg of gabapentin and 1,000 mg of acetaminophen orally. Intraoperatively, patients will receive 4 mg of ondansetron and 15 mg of ketorolac intravenously. Postoperatively, patients will remain on an oral regimen of 300 mg of gabapentin three times daily for one week, and 1,000 mg of acetaminophen and 10 mg of ketorolac every 8 hours for 48 hours after surgery. Additional intraoperative or postoperative opioid analgesics will be administered as needed. Patients with a history of PONV or otherwise deemed high risk for PONV by the attending anesthesiologist will receive a scopolamine patch before induction of general anesthesia.

Data Collection:

Basic demographic data (age, gender, ethnicity) and associated diagnoses such as depression and anxiety will be collected preoperatively. A QoR-15 will be assessed at 24 and 48 hours and 1 week after surgery. Patients will also be sent home with a pain diary to determine pain scores and the amount of pain pills taken for 72 hours after surgery. Other data to be collected will include PACU length of stay and any PACU medications (particularly opioids and rescue antiemetics) given. Opioids will be converted to morphine equivalent doses. The research assistant collecting data will be blinded to the nature of the group assignments.

Study Duration:

We plan to begin enrollment pending IRB approval. The length of participation for each patient will be 1-week in total after surgery.

Statistical Analysis:

Statistical analyses will be performed using STATA 15 statistical software (College Station, TX). Demographic or other categorical data will be analyzed using student's T test or Fisher's exact test as appropriate. Repeated measurements (QoR-15 scores, pain scores) will be analyzed by repeated measures ANOVA or ANOVA on ranks, with further paired comparisons at each time interval performed using the t-test or Mann-Whitney U-test as appropriate. Normally distributed data will be presented as means ± SE of the mean (SEM), non-normally distributed data will be presented as medians ± quartiles (interquartile range) and categorical data will be presented as raw data and as frequencies. The alpha level for all analyses will be set as P<0.05.

Sample size:

Average QOR-15 scores at time point of 24hrs is 112 ± 19 Myles 2016 . A clinically meaningful differences in the QOR-15 scale is 8.0.Myles 2016 Our sample size calculation to detect a 8-point difference in the QOR-15 scale (p<0.05) is 71 patients in each group (alpha=0.05, power=80%). We will inflate our sample size by 10% to account for any missing data or any withdrawal from the study; therefore, our estimated sample size will be 78 patients per group for a total number of patients of 156. Statistical analyses will be performed using STATA 13 statistical software (Dallas, TX).

ELIGIBILITY:
Inclusion Criteria:

* physical ASA status I-III
* age greater than 18 years
* mental competency
* ability to provide informed consent for the study.

Exclusion Criteria:

* severe pulmonary disease including chronic obstructive pulmonary disease(COPD)
* home oxygen use
* a preexisting chronic pain syndrome (defined as daily opioid intake for more than three months prior to surgery)
* allergies to any of the study medications or any of the medications in the multimodal analgesic regimen
* an inability to receive a nerve block due to anticoagulation status infection
* nerve injury
* patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery | 48 Hours
  The primary outcome will be defined as the Quality of Recovery (QoR-15) score at 48 hours after surgery. There are 15 questions assessed on a scale of 0-10, 10 being the better outcome.

SECONDARY OUTCOMES:
Quality of Recovery | 24 hours
  The secondary outcome will be defined as the Quality of Recovery (QoR-15) score at 24 hours after surgery. There are 15 questions assessed on a scale of 0-10, 10 being the better outcome.
Quality of Recovery | 1 Week
  The secondary outcome will be defined as the Quality of Recovery (QoR-15) score at 1 week after surgery. There are 15 questions assessed on a scale of 0-10, 10 being the better outcome.
Pain scores | 72 hours
  Patient reported pain scores on a scale of 0(no pain)-10(extreme pain),
Opioid Use | 72 hours
  Patient reported opioid use for 72 hours.
PACU LOS | 1 Day
  PACU length of stay
PACU Medications | 1 Day
  Measurement of opioid given to patient at PACU in morphine equivalents.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil M Elkassabany, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warrender WJ, Syed UAM, Hammoud S, Emper W, Ciccotti MG, Abboud JA, Freedman KB. Pain Management After Outpatient Shoulder Arthroscopy: A Systematic Review of Randomized Controlled Trials. Am J Sports Med. 2017 Jun;45(7):1676-1686. doi: 10.1177/0363546516667906. Epub 2016 Oct 13. PMID 27729319
- [Background] Uquillas CA, Capogna BM, Rossy WH, Mahure SA, Rokito AS. Postoperative pain control after arthroscopic rotator cuff repair. J Shoulder Elbow Surg. 2016 Jul;25(7):1204-13. doi: 10.1016/j.jse.2016.01.026. Epub 2016 Apr 11. PMID 27079219
- [Background] Hughes MS, Matava MJ, Wright RW, Brophy RH, Smith MV. Interscalene brachial plexus block for arthroscopic shoulder surgery: a systematic review. J Bone Joint Surg Am. 2013 Jul 17;95(14):1318-24. doi: 10.2106/JBJS.L.01116. No abstract available. PMID 23864181
- [Background] Pehora C, Pearson AM, Kaushal A, Crawford MW, Johnston B. Dexamethasone as an adjuvant to peripheral nerve block. Cochrane Database Syst Rev. 2017 Nov 9;11(11):CD011770. doi: 10.1002/14651858.CD011770.pub2. PMID 29121400
- [Background] Kahn RL, Cheng J, Gadulov Y, Fields KG, YaDeau JT, Gulotta LV. Perineural Low-Dose Dexamethasone Prolongs Interscalene Block Analgesia With Bupivacaine Compared With Systemic Dexamethasone: A Randomized Trial. Reg Anesth Pain Med. 2018 Aug;43(6):572-579. doi: 10.1097/AAP.0000000000000817. PMID 29889698
- [Background] Holland D, Amadeo RJJ, Wolfe S, Girling L, Funk F, Collister M, Czaplinski E, Ferguson C, Leiter J, Old J, MacDonald P, Dufault B, Mutter TC. Effect of dexamethasone dose and route on the duration of interscalene brachial plexus block for outpatient arthroscopic shoulder surgery: a randomized controlled trial. Can J Anaesth. 2018 Jan;65(1):34-45. doi: 10.1007/s12630-017-0989-7. Epub 2017 Nov 10. PMID 29127558
- [Background] Tandoc MN, Fan L, Kolesnikov S, Kruglov A, Nader ND. Adjuvant dexamethasone with bupivacaine prolongs the duration of interscalene block: a prospective randomized trial. J Anesth. 2011 Oct;25(5):704-9. doi: 10.1007/s00540-011-1180-x. Epub 2011 Jun 17. PMID 21681533
- [Background] Balocco AL, Van Zundert PGE, Gan SS, Gan TJ, Hadzic A. Extended release bupivacaine formulations for postoperative analgesia: an update. Curr Opin Anaesthesiol. 2018 Oct;31(5):636-642. doi: 10.1097/ACO.0000000000000648. PMID 30074492
- [Background] Viscusi ER. Liposomal drug delivery for postoperative pain management. Reg Anesth Pain Med. 2005 Sep-Oct;30(5):491-6. doi: 10.1016/j.rapm.2005.05.001. No abstract available. PMID 16135355
- [Background] Bowyer A, Jakobsson J, Ljungqvist O, Royse C. A review of the scope and measurement of postoperative quality of recovery. Anaesthesia. 2014 Nov;69(11):1266-78. doi: 10.1111/anae.12730. Epub 2014 Jun 2. PMID 24888412
- [Background] Myles PS. Measuring quality of recovery in perioperative clinical trials. Curr Opin Anaesthesiol. 2018 Aug;31(4):396-401. doi: 10.1097/ACO.0000000000000612. PMID 29846193
- [Background] Chazapis M, Walker EM, Rooms MA, Kamming D, Moonesinghe SR. Measuring quality of recovery-15 after day case surgery. Br J Anaesth. 2016 Feb;116(2):241-8. doi: 10.1093/bja/aev413. PMID 26787793
- [Background] Myles PS, Hunt JO, Nightingale CE, Fletcher H, Beh T, Tanil D, Nagy A, Rubinstein A, Ponsford JL. Development and psychometric testing of a quality of recovery score after general anesthesia and surgery in adults. Anesth Analg. 1999 Jan;88(1):83-90. doi: 10.1097/00000539-199901000-00016. PMID 9895071
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Myles PS, Reeves MD, Anderson H, Weeks AM. Measurement of quality of recovery in 5672 patients after anaesthesia and surgery. Anaesth Intensive Care. 2000 Jun;28(3):276-80. doi: 10.1177/0310057X0002800304. PMID 10853209
- [Background] Myles PS, Myles DB, Galagher W, Chew C, MacDonald N, Dennis A. Minimal Clinically Important Difference for Three Quality of Recovery Scales. Anesthesiology. 2016 Jul;125(1):39-45. doi: 10.1097/ALN.0000000000001158. PMID 27159009